CLINICAL TRIAL: NCT04213547
Title: Sleep Duration and Glycemic Control in Adolescents With Type 2 Diabetes Mellitus
Brief Title: Sleep and Glycemic Control in Type 2 Diabetes Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-016599; 2T32DK063688-16 (NIH)
Record Dates: First submitted 2019-12-26; First posted 2019-12-30 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Aim 2 will be an interventional study design utilizing Fitbit to perform a loss-framed incentive intervention designed to motivate participants to increase their sleep duration with text message feedback. Glycemic control will be measured via laboratory testing of hemoglobin A1c and Libre continuous glucose monitoring (CGM) for 2 weeks pre- and post-intervention.
  A focus group will be conducted prior to this intervention with patients ineligible for the intervention in order to determine appropriate text messaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This will be a single-arm study utilizing a loss-framed incentive intervention to induce increased sleep duration.
  Interventions: Behavioral: Loss frame sleep extension intervention

INTERVENTIONS:
Behavioral: Loss frame sleep extension intervention — Aim 2 will be an interventional study design utilizing Fitbit and text messaging to perform a loss-framed incentive intervention designed to motivate participants to increase their sleep duration. Glycemic control will be measured via laboratory testing of hemoglobin A1c and Libre continuous glucose monitoring (CGM) for 2 weeks pre- and post-intervention. A focus group will be conducted prior to this intervention with patients ineligible for the intervention in order to determine appropriate text messaging.

SUMMARY:
The primary objective is to determine the cross-sectional relationship between sleep duration (as measured by 14 days of actigraphy) and glycemic control in an adolescent Type 2 Diabetes (T2DM) cohort (age 12-20y, n=67). A secondary objective is to determine if a loss-framed incentive for achieving sleep goals can increase sleep duration in 15 adolescent patients diagnosed with T2DM with insufficient sleep. Another secondary objective is to test if increasing sleep duration leads to improved glycemic control in 15 adolescents with T2DM identified in Aim 1 as having <8 hr sleep/evening. A focus group will be conducted prior to this intervention with patients ineligible for the intervention in order to determine appropriate text messaging.

DETAILED DESCRIPTION:
Aim 1 will be a cross-sectional study design utilizing actigraphy watch devices to estimate sleep duration. Participants will be recruited either before or after a routine outpatient clinic visit and asked to complete intake questionnaires. They will then be provided an actigraphy watch device which will be worn for 14 days to estimate sleep duration, and Libre continuous glucose monitor (CGM) to estimate glycemic control. After their visit, clinical data will be extracted from the electronic medical record.

Aim 2 will be an interventional study design utilizing Fitbit to perform a loss-framed incentive intervention designed to motivate participants to increase their sleep duration. Glycemic control will be measured via laboratory testing of hemoglobin A1c and Libre continuous glucose monitoring (CGM) for 2 weeks pre- and post-intervention.

A focus group will be conducted prior to this intervention with patients ineligible for the intervention in order to determine appropriate text messaging.

ELIGIBILITY:
Inclusion Criteria:

Aim 1 for child:

1. Subjects age 12-20
2. Diagnosed with T2DM by standard laboratory criteria without pancreatic autoimmunity
3. Low probability of obstructive sleep apnea (OSA) assessed via validated sleep survey
4. Subjects will be included if they are taking T2DM treatments (i.e., diet modification, Metformin and/or insulin)
5. Parental/guardian permission and child assent

Aim 1 for parent:

1. Parent or legal guardian of child that meets inclusion criteria for Aim 1.

Aim 2 for child:

1. Completed Aim 1 evaluation
2. Average sleep duration < 8 hours per night as determined by actigraphy in Aim 1
3. HbA1c ≤ 10% as HbA1c >10 correlates to poor adherence
4. Adherence > 80%

Focus group for child:

1. Subjects aged 12-20
2. Diagnosed with type 2 diabetes without pancreatic autoimmunity

Exclusion Criteria:

Aim 1 for child:

1. Non-English speaking subject (as questionnaires used are validated in English)
2. Institutionalized patients as sleep duration will not be of their own accord, and therefore is not generalizable to the rest of the adolescent T2DM population.
3. Patients with other forms of Diabetes Mellitus (e.g. Type 1 Diabetes)
4. Behavioral disorders that may affect data collection (e.g. autism spectrum disorder) will be determined on a case-by-case basis. These include patients that are unable to answer questionnaires on their own, participate in a sleep diary, wear devices and/or understand incentives.
5. Oral or IV steroid treatment within the past month
6. Females with known pregnancies as these patients will not be generalizable to the rest of the adolescent T2DM population and pregnancy may alter sleep duration.
7. Subjects with known hyperthyroidism, pain syndrome, or serious medical condition that can affect sleep.
8. Subjects with hemoglobinopathies that affect hemoglobin A1c measurement.
9. Unable to obtain point-of-care hemoglobin A1c in clinic on date of recruitment
10. Known diagnosis of obstructive sleep apnea or other sleep disorder

Aim 1 for Parent:

1. Non-English speaking subject (as questionnaires used are validated in English)
2. Parent/guardians with cognitive disorders that may affect data collection (determined on a case-by-case basis)

Aim 2 for child:

1. Do not own a smart phone or tablet

Focus group for child:

1. Non-English speaking subject (as focus group will be conducted in English)
2. Lack of access to a computer, tablet or smartphone that can accommodate participation in video conferencing

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Sleep duration (for Aim 2) | 13 weeks
  Will assess for sleep extension throughout intervention
Hemoglobin A1c (for Aim 1) | baseline
  Aim 1 is assessing cross-sectional relationship of A1c to sleep duration
BMI (for Aim 1) | baseline
  Aim 1 is assessing cross-sectional relationship of BMI to sleep duration
Qualitative data from focus group | baseline at focus group
  Qualitative output from focus group discussion on text messages

SECONDARY OUTCOMES:
Glycemic control | 13 weeks
  Will assess for change in hemoglobin a1c throughout intervention
Glycemic control | 13 weeks
  Will assess for change in continuous glucose monitor measures throughout intervention
BMI | 13 weeks
  Will assess for change in body mass index (BMI) throughout intervention

CONTACTS AND LOCATIONS:
Overall Officials: Talia A Hitt, MD/MPH, Study Director — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mayer-Davis EJ, Lawrence JM, Dabelea D, Divers J, Isom S, Dolan L, Imperatore G, Linder B, Marcovina S, Pettitt DJ, Pihoker C, Saydah S, Wagenknecht L; SEARCH for Diabetes in Youth Study. Incidence Trends of Type 1 and Type 2 Diabetes among Youths, 2002-2012. N Engl J Med. 2017 Apr 13;376(15):1419-1429. doi: 10.1056/NEJMoa1610187. PMID 28402773
- [Background] Cappuccio FP, Taggart FM, Kandala NB, Currie A, Peile E, Stranges S, Miller MA. Meta-analysis of short sleep duration and obesity in children and adults. Sleep. 2008 May;31(5):619-26. doi: 10.1093/sleep/31.5.619. PMID 18517032
- [Background] Wheaton AG, Olsen EO, Miller GF, Croft JB. Sleep Duration and Injury-Related Risk Behaviors Among High School Students--United States, 2007-2013. MMWR Morb Mortal Wkly Rep. 2016 Apr 8;65(13):337-41. doi: 10.15585/mmwr.mm6513a1. PMID 27054407
- [Background] Buxton OM, Pavlova M, Reid EW, Wang W, Simonson DC, Adler GK. Sleep restriction for 1 week reduces insulin sensitivity in healthy men. Diabetes. 2010 Sep;59(9):2126-33. doi: 10.2337/db09-0699. Epub 2010 Jun 28. PMID 20585000
- [Background] Spiegel K, Knutson K, Leproult R, Tasali E, Van Cauter E. Sleep loss: a novel risk factor for insulin resistance and Type 2 diabetes. J Appl Physiol (1985). 2005 Nov;99(5):2008-19. doi: 10.1152/japplphysiol.00660.2005. PMID 16227462
- [Background] Knutson KL, Van Cauter E, Zee P, Liu K, Lauderdale DS. Cross-sectional associations between measures of sleep and markers of glucose metabolism among subjects with and without diabetes: the Coronary Artery Risk Development in Young Adults (CARDIA) Sleep Study. Diabetes Care. 2011 May;34(5):1171-6. doi: 10.2337/dc10-1962. Epub 2011 Mar 16. PMID 21411507
- [Background] Patel MS, Asch DA, Rosin R, Small DS, Bellamy SL, Heuer J, Sproat S, Hyson C, Haff N, Lee SM, Wesby L, Hoffer K, Shuttleworth D, Taylor DH, Hilbert V, Zhu J, Yang L, Wang X, Volpp KG. Framing Financial Incentives to Increase Physical Activity Among Overweight and Obese Adults: A Randomized, Controlled Trial. Ann Intern Med. 2016 Mar 15;164(6):385-94. doi: 10.7326/M15-1635. Epub 2016 Feb 16. PMID 26881417